CLINICAL TRIAL: NCT02035371
Title: A Trial Investigating the Pharmacokinetic Properties of FIAsp in Children, Adolescents and Adults With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1218-3888; 2011-002104-32 (EudraCT Number); U1111-1121-1469 (Other: WHO)
Record Dates: First submitted 2014-01-10; First posted 2014-01-14 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FIAsp (Experimental): Each subject will be randomly allocated to a treatment sequence consisting of 2 dosing visits separated by a wash-out period of 3-12 days
  Interventions: Drug: Faster-acting insulin aspart
- NovoRapid® (Active Comparator): Each subject will be randomly allocated to a treatment sequence consisting of 2 dosing visits separated by a wash-out period of 3-12 days
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: Faster-acting insulin aspart — A single dose will be administered subcutaneously (s.c. under the skin)
  Arms: FIAsp
Drug: insulin aspart — A single dose will be administered subcutaneously (s.c. under the skin)
  Arms: NovoRapid®

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the pharmacokinetic (the exposure of the trial drug in the body) properties of FIAsp (faster-acting insulin aspart) in children, adolescents and adults with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 6-64 years (both inclusive) at the time of signing informed consent
* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Body mass index (BMI) for children and adolescents (male and female) between the 3rd and 97th BMI percentile and for adults equal to or below 28.0 kg/m^2

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking at least one cigarette, cigar or pipe daily)
* Not able or willing to refrain from smoking and use of nicotine substitute products during the inpatient period

Ages: 6 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2014-01-13 (Actual); Primary Completion 2014-07-24 (Actual); Study Completion 2014-07-24 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin aspart concentration-time curve | From 0 to 12 hours

SECONDARY OUTCOMES:
Maximum observed serum insulin aspart concentration | From 0-12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Hanover, Germany

REFERENCES:
- [Background] Danne T, Biester T, Fath M, Thorsson L, Rikte T, Kordonouri O, Haahr H. Earlier onset and higher early exposure of faster-acting insulin aspart vs. insulin aspart in adults is retained in children and adolescents with T1D. Diabetes 2015; 64 (Suppl. 1): A247 (976-P)
- [Background] Heise T, Pieber TR, Danne T, Erichsen L, Haahr H. Faster Onset and Greater Early Exposure and Glucose-Lowering Effect with Faster-Acting Insulin Aspart vs. Insulin Aspart: A Pooled Analysis in Subjects with Type 1 Diabetes. Diabetes. 2016; Suppl. 1: A239. doi:10.2337/db16-861-1374 http://dx.doi.org/10.2337/db16-861-1374
- [Result] Fath M, Danne T, Biester T, Erichsen L, Kordonouri O, Haahr H. Faster-acting insulin aspart provides faster onset and greater early exposure vs insulin aspart in children and adolescents with type 1 diabetes mellitus. Pediatr Diabetes. 2017 Dec;18(8):903-910. doi: 10.1111/pedi.12506. Epub 2017 Feb 6. PMID 28165180
- [Derived] Heise T, Pieber TR, Danne T, Erichsen L, Haahr H. A Pooled Analysis of Clinical Pharmacology Trials Investigating the Pharmacokinetic and Pharmacodynamic Characteristics of Fast-Acting Insulin Aspart in Adults with Type 1 Diabetes. Clin Pharmacokinet. 2017 May;56(5):551-559. doi: 10.1007/s40262-017-0514-8. PMID 28205039
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com